CLINICAL TRIAL: NCT01386372
Title: A Pilot Study To Evaluate The Incidence Of Hyponatremia In A Medical-Surgical Hospital And To Explore The Efficacy And Safety Of Tolvaptan In The Clinical Practice
Brief Title: Tolvaptan for In-hospital Hyponatremia
Acronym: INSERT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INSERT; 2010-024431-17 (EudraCT Number)
Record Dates: First submitted 2011-06-24; First posted 2011-07-01 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2013-02

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Vasopressin; Tolvaptan; SIADH
MeSH Terms: conditions — Hyponatremia; Diabetes Insipidus; Inappropriate ADH Syndrome | interventions — Tolvaptan; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tolvaptan (Experimental)
  Interventions: Drug: Tolvaptan
- standard therapy (Active Comparator)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: Tolvaptan — Patients will receive full-dose oral tolvaptan therapy up to 1 month after randomization. During the initial 4 days of therapy, the dose of the study drug will be increased from 15 to 30 mg or from 30 to 60 mg according to a regimen designed for slow correction of serum sodium concentrations to 135 mEq/L or more Depending on the serum sodium concentration the dose will be increased or decreased. Patients will then be continued on their maintenance therapy with adjustments allowed to prevent hyponatremia and avoiding hypernatremia. As soon as normal serum sodium levels are achieved in at least two consecutive measurements the dose of the study drug will be progressively tapered according to an individually tailored weaning program
  Arms: Tolvaptan
Other: Standard therapy — Fluid restriction, normal or hypertonic saline, furosemide.
  Arms: standard therapy

SUMMARY:
Hyponatremia is a common electrolyte disorder encountered in hospitalized patients. A preliminary, observational, feasibility analysis finalized to assess retrospectively the incidence of hyponatremia (Serum sodium < 135 mEq/L) in a general medical-surgical hospital and the distribution of the cases of hyponatremia among different referral units showed that over one year observation there were more than 1500 cases of hyponatremia. Conventional therapy for hyponatremia depends on its causes, speed of onset, extracellular fluid volume status, and severity. Treatment consists in fluid restriction, normal or hypertonic saline, furosemide. Recent development of arginine vasopressin antagonists has provided a new therapeutic option for treatment of hyponatremia.Tolvaptan, an orally administered, nonpeptide, selective vasopressin V2 receptor antagonist reported to increase free water clearance and limit fluid retention in subjects with congestive heart failure or liver cirrhosis, has been also shown to be effective in the treatment of chronic hyponatremia in patients with SIADH, chronic heart failure, liver cirrhosis. Thus the investigators designed a clinical study to explore the incidence of severe hyponatremia in hospitalized patients in the setting of large general hospital and to evaluate whether tolvaptan is effective and safe in increasing serum sodium concentration in patients with normovolemic and hypervolemic hyponatremia in the setting of daily clinical practice. Moreover this study may help understand the cost-effectiveness of tolvaptan therapy compared to traditional treatments of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Non artifactual hyponatremia in euvolemic or hypervolemic states, defined as serum sodium <135 mEq/L confirmed in at least 2 consecutive evaluations;
* 18 years of age or older;
* Able to give written Informed Consent.

Exclusion Criteria:

* Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods;
* Hyponatremia in hypovolemic states;
* Acute and transient hyponatremia associated with head trauma or post-operative state;
* Hyponatremia due to uncontrolled hypothyroidism or uncontrolled adrenal insufficiency;
* Cardiac surgery within 30 days prior to the potential study enrollment, excluding percutaneous coronary interventions;
* History of a myocardial infarction within 30 days prior to the potential study enrollment;
* History of sustained ventricular tachycardia or ventricular fibrillation within the last 30 days, unless in the presence of an automatic implantable cardioverter defibrillator;
* Severe angina including angina at rest or at slight exertion and/or unstable angina;
* History of a cerebrovascular accident within the last 30 days;
* Subjects with psychogenic polydipsia may not be included, however subjects with other psychiatric illness may be included;
* Systolic arterial blood pressure <90 mmHg;
* History of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benazepril);
* History of drug or medication abuse within the past year, or current alcohol abuse;
* Uncontrolled diabetes mellitus defined as fasting glucose >300mg/dL;
* Urinary tract obstruction except BPH if non-obstructive;
* Terminally ill or moribund condition with little chance of short-term survival;
* Serum creatinine >3.5 mg/dL;
* Serum sodium <120 mEq/L with associated neurologic impairment, i.e. symptoms such as apathy, confusion, seizures;
* Patients with progressive or episodic neurologic disease such as multiple sclerosis or history of multiple strokes;
* Child-Pugh score greater than 10 (unless approved);
* Patients receiving intravenous fluids at a rate greater than KVO (Keep Vein Open);
* Hyponatremia due to lab artifacts;
* Patients receiving AVP or its analogs for treatment of any condition;
* Patients receiving within 7 days of randomization, other medications for treatment of hyponatremia specifically: demeclocycline, lithium carbonate or urea;
* Patients likely requiring IV saline for correction of symptomatic or asymptomatic severe hyponatremia during the course of the study;
* Severe pulmonary artery hypertension;
* Hyponatremia should not be the result of any medication that can safely be withdrawn.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in proportion of subjects with normonatremia at 6 month. | At 1,2,3,4 and 10 day, and at 1,2,4 and 6 month..
Changes from baseline in serum sodium levels from basal at 6 months. | At 1,2,3,4, 10 day and at 1,2,4 and 6 month..

SECONDARY OUTCOMES:
Proportion of subjects achieving normonatremia at discharge and at predefined time-points. | 8 hours, 1, 2, 3, and 10 days and 1, 2, 4 and 6 months after randomization
Absolute changes in serum sodium levels vs baseline at predefined time-points. | 8 hours, 1, 2, 3, and 10 days and 1, 2, 4 and 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- OO.RR., Bergamo - Unit of Nephrology and Dialisis, Bergamo, Italy